CLINICAL TRIAL: NCT00706693
Title: The Effectiveness of Glucose, Sucrose and Fructose in Treating Hypoglycemia in Children With Type 1 Diabetes
Brief Title: Skittles(TM) Effective for Treating Hypoglycemia in Children With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Canadian Diabetes Association (Other); LifeScan Canada (Unknown); Becton, Dickinson and Company (Industry)
Responsible Party: Allison Husband, RN, MN, CDE, Alberta Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 17089-AH
Record Dates: First submitted 2008-06-25; First posted 2008-06-27 (Estimated); Last update posted 2008-07-09 (Estimated); Status verified 2008-07

CONDITIONS: Type 1 Diabetes Mellitus; Hypoglycemia
Keywords: hypoglycemia; treatment; glucose; sucrose; fructose
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Glucose (Active Comparator): BD glucose tablets (TM) are taken PO in response to a hypoglycemic event by participants randomized to this arm
  Interventions: Dietary Supplement: Ingestion of BD glucose tablets (TM)
- Fructose (Active Comparator): Fruit to Go (TM) is taken PO in response to a hypoglycemic event by participants randomized to this arm
  Interventions: Dietary Supplement: Ingestion of Fruit to Go (TM)
- Sucrose (Active Comparator): Skittles (TM) are taken PO in response to a hypoglycemic event by participants randomized to this arm
  Interventions: Dietary Supplement: Ingestion of Skittles (TM)

INTERVENTIONS:
Dietary Supplement: Ingestion of BD glucose tablets (TM) — Hypoglycemia (blood glucose is less than 4.0 mmol/L as measured by a glucose meter) will be treated with BD glucose tablets by giving 10g of glucose in children 10 and under. Children and teens over 10 will receive 15g of glucose.
  Arms: Glucose
Dietary Supplement: Ingestion of Skittles (TM) — Hypoglycemia (blood glucose is less than 4.0 mmol/L as measured by a glucose meter) will be treated with Skittle by giving 10g of sucrose in children 10 and under. Children and teens over 10 will receive 15g of sucrose.
  Arms: Sucrose
Dietary Supplement: Ingestion of Fruit to Go (TM) — Hypoglycemia (blood glucose is less than 4.0 mmol/L as measured by a glucose meter) will be treated with Fruit to Go by giving 10g of fructose in children 10 and under. Children and teens over 10 will receive 15g of fructose.
  Arms: Fructose

SUMMARY:
The purpose of this study is to determine the most effective treatment option for managing naturally occurring hypoglycemia in children with type 1 diabetes.

Hypotheses:

1. Sucrose and Fructose are equally effective as glucose in the treatment of spontaneous hypoglycemia in children with type 1 diabetes.
2. Children and teens will use a variety of treatment practices for the management of hypoglycemia.
3. Children and teens will prefer the mode of treatment that was most effective in treating hypoglycemia.

DETAILED DESCRIPTION:
An open labeled, randomized, cross-over design will be used. Each subject will treat 5 hypoglycemic events with glucose, 5 with sucrose and 5 with fructose. Subjects will be randomized into order of treatment.

Primary Objective:

1. To determine if sucrose and fructose are equally effective as glucose in the treatment of spontaneous hypoglycemia in children with type 1 diabetes.

   Secondary Objectives:
2. To determine present hypoglycemia treatment practices of children and teens with type 1 diabetes (prior to entry into the study).
3. To determine preferred mode of treatment for hypoglycemia after completing the study.

Inclusion Criteria:

The sample will consist of 65 individuals with a history of type 1 diabetes (based on clinical presentation) for three or more months and who are between the ages of 3 and 18 years. All eligible participants will be patients of the Alberta Children's Hospital Diabetes Clinic.

Exclusion Criteria:

Individuals with the following conditions/circumstances will be excluded from the study:

* adrenal insufficiency
* uncompensated hypothyroidism
* clinical autonomic neuropathy
* celiac disease
* lack of family support
* unwilling or unable to follow the study protocol
* subjects with less than 4 hypoglycemic events per month

Instruments:

Blood glucose will be measured with a blood glucose meter. All meters will have a lab to meter comparison performed. In accordance with the 1998 Clinical Practice Guidelines for Diabetes Management in Canada, an acceptable meter value will be +15% of the lab value (7). Participants will be provided with a complimentary meter and strips.

All participants will be provided with a digital timer to enable accurate 15 minute timing of post treatment blood glucose.

A Demographic and Pre-Study Data tool has been developed to collect pre-study information (see Appendix B) as well as a Low Blood Glucose Treatment Log to record pre- and post-treatment blood glucose results (see Appendix C).

Study Procedure:

A letter inviting participation in the study will be mailed to all eligible participants (see Appendix D). Further recruitment will be done during clinic appointments. Six months will be allocated for recruitment of subjects. Subjects will meet with the study research assistant and informed and signed consent will be obtained. Participants will be assigned a study number based on their order of recruitment. The research assistant and participant will not determine treatment order. Each participant will be assigned a treatment order based on a randomization table (See Table 1).

The research assistant will also obtain demographic data and information on present hypoglycemia treatment practices, explain the study protocol, and provide Study Protocol instructions (see Appendix E). The lab/meter comparison will be obtained prior to data collection.

The study protocol is as follows:

* Hypoglycemia will be confirmed with a blood glucose test.
* If blood glucose is less than 4.0 mmol/L it will be treated with pre-packaged treatments and in the order determined by randomization.
* The blood glucose will be re-tested 15 minutes after treatment.
* If the blood glucose is still less than 4.0 mmol/L, it will be treated again as per study protocol and then re-tested 15 minutes later.
* If the next meal or snack is more than 1 hour away, a snack containing 15 g of carbohydrate and a protein will be eaten.
* Participants will record blood glucose results and treatment method on the Low Blood Glucose Treatment Log.

If participants can not follow the above outlined protocol, they will be instructed to treat as per usual practice and not record data. This will mean that most hypoglycemic events treated as per protocol will likely occur when children are with their parents or in the comfort of their own homes.

Assuming that children and teens will experience 1 to 3 hypoglycemic events per week, it is anticipated that data collection will occur over a 5 to 15 week period. The research assistant will call participants every two weeks to monitor study progress. Once the subject has treated 15 hypoglycemic episodes as per study protocol and completed the Low Blood Glucose Treatment Log, they will return it in a pre-addressed and stamped envelope. There will be a question at the end of the Low Blood Glucose Treatment Log asking preferred method of hypoglycemia treatment following completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus
* Diagnosed 6 or more months ago
* Patient of the Alberta Children's Hospital Diabetes Clinic

Exclusion Criteria:

* Adrenal insufficiency
* Uncompensated hypothyroidism
* Clinical autonomic neuropathy
* Celiac disease
* Lack of family support
* Unwilling or unable to follow the study protocol
* Subjects with less than 4 hypoglycemic events per month

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2003-08; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
To determine if sucrose and fructose are equally effective as glucose in the treatment of spontaneous hypoglycemia in children with type 1 diabetes. | 15 minutes

SECONDARY OUTCOMES:
To determine present hypoglycemia treatment practices of children and teens with type 1 diabetes (prior to entry into the study).
To determine preferred mode of treatment for hypoglycemia after completing the study.

CONTACTS AND LOCATIONS:
Overall Officials: Allison Husband, RN, MN, CDE, Principal Investigator — Alberta Children's Hospital
Locations (1):
- Alberta Children's Hospital, Calgary, Alberta, Canada

REFERENCES:
- [Result] Husband AC, Crawford S, McCoy LA, Pacaud D. The effectiveness of glucose, sucrose, and fructose in treating hypoglycemia in children with type 1 diabetes. Pediatr Diabetes. 2010 May;11(3):154-8. doi: 10.1111/j.1399-5448.2009.00558.x. Epub 2009 Aug 3. PMID 19663922